CLINICAL TRIAL: NCT02098057
Title: A Pilot Study Barrier Function, Intestinal Permeability and Tight Junction Expression in Gluten Sensitive Patients With Functional Gastrointestinal Disorders
Brief Title: Change in Permeability of the Small Intestine After Treatment With Gluten
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria I. Vazquez Roque, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 13-005160; FP00074933 (Other: CRT-1)
Record Dates: First submitted 2014-03-14; First posted 2014-03-27 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Gastrointestinal Disorders
Keywords: IBS-diarrhea
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): A total of 24 patients with NCGS and 12 healthy controls will be recruited for this study. The 24 patients with NCGS will be randomized to receive one of two diets (GFD or GCD) in a 1:1 ratio
  Interventions: Drug: Placebo
- Gluten (Active Comparator): A total of 24 patients with NCGS and 12 healthy controls will be recruited for this study. The 24 patients with NCGS will be randomized to receive one of two diets (GFD or GCD) in a 1:1 ratio
  Interventions: Dietary Supplement: Gluten Healthy

INTERVENTIONS:
Dietary Supplement: Gluten Healthy — Assessment of current diet and amount of gluten consumed will be determined by the dietitian and by means of a questionnaire at baseline. Subjects will have a 2-week run in period, in which they will continue or initiate a gluten free diet plan prepared by the dietitians. After the run-in period, participants will be randomized to either a gluten containing diet (GCD) or placebo (GFD) for 4 weeks.
  Arms: Gluten
Drug: Placebo — A total of 24 patients with NCGS and 12 healthy controls will be recruited for this study. The 24 patients with NCGS will be randomized to receive one of two diets (GFD or GCD) in a 1:1 ratio
  Assessment of current diet and amount of gluten consumed will be determined by the dietitian and by means of a questionnaire at baseline. Subjects will have a 2-week run in period, in which they will continue or initiate a gluten free diet plan prepared by the dietitians. After the run-in period, participants will be randomized to either a gluten containing diet (GCD) or placebo (GFD) for 4 weeks.
  Arms: Placebo

SUMMARY:
The overall hypothesis of this research study is that gluten intake alters intestinal barrier function in patients with Irritable Bowel Syndrome (IBS) diarrhea who also exhibit non-celiac gluten sensitivity (NCGS).

DETAILED DESCRIPTION:
The specific aim of this hypothesis-generating, pilot study is to randomize (like the flip of a coin) patients who have Non Celiac Gluten Sensitivity to a 4-week Gluten-containing diet (GCD) or to a Gluten free diet (GFD). The study will evaluate small bowel (SB) permeability functionally (2-sugar differential excretion), morphologically, using probe-based confocal laser to evaluate the small intestinal, as well as molecularly, using tight junction (TJ) messenger RNA (mRNA) expression in small bowel mucosa in response to the different diets.

ELIGIBILITY:
Inclusion Criteria:

1. Non celiac gluten sensitive patients with a functional bowel disorder
2. Age 18 to 70 years.

Exclusion Criteria:

1. Positive serum tissue transglutaminase (TTG) Immunoglobulin A (IgA) positive or medical record of small bowel biopsy suggestive of celiac disease.
2. Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability).
3. Abdominal surgeries (except appendectomy, cholecystectomy and vaginal hysterectomy or tubal ligation)
4. Use of Nonsteroidal Anti-inflammatory Drugs(NSAIDs) or aspirin within the past week (since Nonsteroidal Anti-inflammatory Drugs (NSAIDs) affect intestinal permeability).
5. Use of oral corticosteroids within the previous 6 weeks.
6. Ingestion of artificial sweeteners such as Sucralose, Nutrasweet ™ (aspartame), lactulose or mannitol 2 days before the study tests begins, e.g., foods to be avoided are sugarless gums or mints and diet soda.
7. Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies.
8. High anxiety or depression score (>11 on each subscale) on the Hospital Anxiety Depression Score questionnaire.
9. Known allergy to fluorescein.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Change in permeability of the small intestine after treatment | Baseline to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Vazquez Roque, MD, MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share Individual Patient Data at this time. Once data analysis is done at study conclusion, it will help determine feasibility for moving forward with another, similar - possibly larger, study. That said, data may be released after study conclusion.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials